CLINICAL TRIAL: NCT03371303
Title: Analysis of Changes in Medication Prescriptions After Hospitalization for 4 Disciplines: Gerontology, Diabetology, Cardiology and Rheumatology: Medical, Pharmaceutical and Economic Aspects
Acronym: PHMEV
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-25
Record Dates: First submitted 2017-12-01; First posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Diabetes; Cardiac Disease; Rheumatic Diseases
MeSH Terms: conditions — Diabetes Mellitus; Heart Diseases; Rheumatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- diabetology
  Interventions: Other: collection of prescription data
- cardiology
  Interventions: Other: collection of prescription data
- rheumatology
  Interventions: Other: collection of prescription data
- geriatrics
  Interventions: Other: collection of prescription data

INTERVENTIONS:
Other: collection of prescription data — collection of prescription data before and after a hospitalization

SUMMARY:
The modifications of the medicinal treatments secondary to the hospitalizations have multiple reasons: reassessment of the previous treatment (conciliation), new therapeutic necessities, potential risk of iatrogeny or of drug interaction, restrictions of the therapeutic booklet, classification in reserve or hospital prescription ... These modifications are potentially generating extra costs for the Health Insurance and are monitored under the terms of the Contract of Good Use. The aims of this analysis are to define the medical-pharmaceutical rationale of the treatment changes imposed by hospitalization in a university-hospital center, their influence on the security of the medical treatment of patients and their financial implications for healthcare organizations

ELIGIBILITY:
inclusion criteria

* Patient social insured
* Patient belonging to the general social security scheme
* Patient followed in cardiology, rheumatology, geriatrics or diabetology departments

no exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients must be hospitalized in one of the services of a university hospital, in the following 4 disciplines: diabetology, geriatrics, cardiology and rheumatology
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
entry orders before hospitalization | 15 months
exit orders after hospitalization | 15 months

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France